CLINICAL TRIAL: NCT03068117
Title: A Multicentre, Non-blinded, Randomised Controlled Trial to Assess the Impact of Regular Early SPEcialist Symptom Control Treatment on Quality of Life in Malignant Mesothelioma - "RESPECT-Meso"
Brief Title: Malignant Mesothelioma - Can we Improve Quality of Life
Acronym: RESPECT-Meso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: British Lung Foundation (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHT/2013/46
Record Dates: First submitted 2017-01-04; First posted 2017-03-01 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Mesothelioma, Malignant
Keywords: Specialist Palliative Care; Symptom Control; Early Referral; Quality of Life; Malignant Pleural Mesothelioma; Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RESSCT plus Standard Care/Therapy (Experimental): Regular Early Specialist Symptom Control Treatment (RESSCT) and Standard Therapy.
  Participants will be seen within three weeks of randomisation by the Specialist Palliative Care Team (SPCT), (regardless of, and in addition to, all other treatments being offered). The initial meeting will be an approximately 1 hour consultation with a member of the Specialist Palliative Care team. This may be either a Consultant or Specialist Palliative Care Clinical Nurse Specialist (SPCCNS).
  Patients will then continue to be seen regularly on at least a 4 weekly basis (regardless of other treatments, interventions and symptoms) by a member of the SPCT, with consultations lasting approximately 30 minutes. These monthly reviews will continue until end of trial (EOT) or patient death.
  Interventions: Other: Regular Early Specialist Symptom Control Treatment (RESSCT)
- Standard Care/Therapy (No Intervention): The standard care/therapy control group will continue to receive all appropriate, standard treatment for Malignant Pleural Mesothelioma (MPM) currently available to them and will be initiated by the patient's General Practitioner (GP), the cancer MDT or lead respiratory physician as required.

INTERVENTIONS:
Other: Regular Early Specialist Symptom Control Treatment (RESSCT) — Participants will be seen within three weeks of randomisation by the Specialist Palliative Care Team (SPCT), (regardless of, and in addition to, all other treatments being offered). The initial meeting will be an approximately 1 hour consultation with a member of the Specialist Palliative Care team. This may be either a Consultant or Specialist Palliative Care Clinical Nurse Specialist (SPCCNS).
  Patients will then continue to be seen regularly on at least a 4 weekly basis (regardless of other treatments, interventions and symptoms) by a member of the SPCT, with consultations lasting approximately 30 minutes. These monthly reviews will continue until end of trial (EOT) or patient death.
  Other Names: Regular Early Specialist Palliative Care
  Arms: RESSCT plus Standard Care/Therapy

SUMMARY:
Patients with malignant pleural mesothelioma (MPM) frequently have significant physical symptoms, with up to 92% of patients complaining of three or more symptoms at presentation. Such symptom scores are similar to those reported in advanced non small cell lung cancer (NSCLC) and have been demonstrated to correlate with interference with activity and worse quality of life (QOL). Several studies have reported that baseline Quality of Life (QOL) is a significant prognostic factor for survival in NSCLC patients. In 2010, a non-blinded randomised controlled trial of 151 patients in the United States (US) demonstrated an improved QOL, fewer depressive symptoms and improved survival with early, regular specialist palliative care team (SPCT) involvement in addition to their routine care.

The RESPECT-Meso study will examine the effect on quality of life following early Specialist Palliative Care (SPC) involvement for Regular Early Symptom Control Treatment (RESSCT) in addition to routine care in patients with newly diagnosed MPM in the United Kingdom (UK).

DETAILED DESCRIPTION:
The purpose of this study is to examine if regular early Specialist Symptom Control Treatment (SSCT) involvement in mesothelioma patients can improve patients' and carers' quality of life (QOL) during their illness.

Mesothelioma is a cancer of the lining around the chest wall which is caused by asbestos exposure. The UK has the highest death rate from mesothelioma in the world and mesothelioma will soon account for approximately 1 in 170 of all deaths in the UK. At present, there is no cure. About a third of patients have chemotherapy, which can prolong how long patients live ('survival') by a few months. For many patients, doctors can only offer treatment of symptoms from the cancer, rather than treating the cancer itself. For most patients, survival is usually between 8-12 months.

Mesothelioma causes many symptoms including breathlessness, chest pain, weight loss and fatigue. Specialist Palliative Care (SPC) medicine doctors and nurses are specialists in treating symptoms due to life limiting illness. They also provide emotional support for patients and carers. The current practice in the UK is to involve SPC towards the end of a patient's life. A recent study from America examining lung cancer patients showed that involving SPC early in a patient's treatment improved patients' QOL during their illness, and also their survival.

Until a cure for, or significant advance in the treatment of, MPM becomes available, attempts to improve the QOL of patients and carers will remain the primary goal of teams managing their care. Recent research examining NSCLC and early SPCT intervention by Temel et al demonstrated that such a novel approach is plausible, possible and effective in improving patients' QOL. This report demonstrated a survival benefit of 2.7 months; if a new chemotherapy drug were to demonstrate such an effect, it would likely be considered a significant breakthrough in the treatment of MPM.

Current practice in the UK is to involve SPC towards the final months, and perhaps weeks, of a life-limiting illness. Therefore, the regular early SSCT intervention is well-placed to demonstrate any effects from the proposed intervention.

This comprehensive, randomised, multicentre study will examine both patient and caregiver QOL, and the healthcare economic consequences of providing such an intervention. The results of such will be widely applicable to many institutions and patients throughout the UK.

This study will randomly divide patients to either all normal treatment and support ('usual care', as is always offered), or usual care and regular SPC consultations from the time of diagnosis. No treatments will be withheld; this study is providing additional support to patients and their families. Patients will be asked to complete a set of questionnaires at the start of the study, and then monthly for up to 6 months. Carers will also complete a set of questionnaires at the start of the study and then at 3 and 6 months. Reported QOL and survival between the two groups will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of malignant pleural mesothelioma (MPM)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1. (Asymptomatic patients score 0; symptomatic but ambulatory patients score 1)
* The diagnosis of MPM received within the last 6 weeks
* Ability to provide written informed consent in English and comply with trial procedures

Exclusion Criteria:

* Other known malignancy within 5 years (excluding localised squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, grade III and low grade prostate cancer (Gleason score <5, with no metastases)).
* Significant morbidity which the lead physician (or MDT) feel will unduly confound or influence QOL.
* Those patients the MDT judge require referral to the SPCT at the point of diagnosis.
* Concurrent, or less than 3 months, since participation in another non-mesothelioma clinical trial that may affect QOL.
* Participation in a concurrent mesothelioma trial, within 12 weeks after randomisation, that may affect QOL.
* Referral at the time of recruitment for cytoreductive, tumour de-bulking, radical decortication or extrapleural pneumonectomy surgery for MPM. (Video Assisted Thoracoscopic Surgery or 'mini' thoracotomy for pleurodesis and diagnosis attempts are permissible.)
* Chemotherapy treatment for MPM initiated prior to consent.
* A significant history of depression / anxiety / psychiatric illness requiring specialist hospital care within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
EORTC C-30 Quality of Life | 12 weeks
  The primary objective of this randomised controlled study is to assess the impact of regular early specialist symptom control treatment (SSCT) involvement on global quality of life (QOL) in patients recently diagnosed with malignant pleural mesothelioma (MPM) 12 weeks post randomisation as compared to standard care.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) in Patients | Baseline & 24 weeks
  The following questionnaire will be used to measure HRQoL in patients;
  - EORTC C-30
  This will be completed at baseline & 24 weeks following randomisation.
Health Related Quality of Life (HRQoL) in Patients | Baseline 12 & 24 weeks
  The following questionnaire will be used to measure HRQoL in patients;
  - EORTC LC-13
  This will be completed at baseline, 12 & 24 weeks following randomisation.
Health Related Quality of Life (HRQoL) in Patients | Baseline, 12 & 24 weeks
  The following questionnaire will be used to measure HRQoL in patients;
  - EuroQol-5 Dimension questionnaire (EQ-5D)
  This will be completed at baseline, 12 & 24 weeks following randomisation.
Patient Mood | Baseline, 12 & 24 weeks
  The following questionnaire will be used to measure mood in patients;
  - Global Health Questionnaire (GHQ) 12
  This will be completed at baseline, 12 & 24 weeks following randomisation.
Primary Caregiver Health Related Quality of Life (HRQoL) | Baseline, 12 & 24 weeks & 24 weeks post mortality of the patient.
  The following questionnaires will be used to measure HRQoL in primary caregivers;
  - Short Form 36 item questionnaire (SF-36)
  This will be completed at baseline, 12 & 24 weeks following randomisation and subsequently at 24 week post patient mortality.
Primary Caregiver Mood | Baseline, 12 & 24 weeks & 24 weeks post mortality of the patient.
  The following questionnaires will be used to measure mood in primary caregivers;
  - Global Health Questionnaire (GHQ) 12
  This will be completed at baseline, 12 & 24 weeks following randomisation and subsequently at 24 week post patient mortality.
Overall Survival between the two study groups | From randomisation to death or end of study (whichever occurs first), assessed up to 38 months
  Overall survival from date of randomisation will be compared. Patients alive at the End of the Study will be recorded as 'alive' to ensure there is no missing data.
Healthcare Utilisation between the two study groups | up to 24 weeks post patients death
  Healthcare resource use will be obtained from hospital, hospice and primary care databases after patient death or End of Study.
Primary caregiver satisfaction with end of life care | 12 & 24 weeks and 24 weeks post mortality
  Primary caregiver satisfaction with end of life care as assessed by the Family Caregive Survey 2 (FAMCARE-2) questionnaire at 12 & 24 weeks and 24 weeks post mortality of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Anoop J Chauhan, PhD, FRCP, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (19):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- United Kingdom (18):
  - County Durham and Darlington NHS Foundation Trust, County Durham, Durham
  - Basildon and Thurrock University Hospitals NHS Foundation Trust - Basildon Hospital, Basildon, Essex
  - Mid Essex Hospital Services NHS Trust - Broomfield Hospital, Chelmsford, Essex
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - Sherwood Forest Hospitals NHS Foundation Trust, Nottingham, Nottinghamshire
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Nottinghamshire
  - Taunton and Somerset NHS Foundation Trust - Musgrove Park Hospital, Taunton, Somerset
  - Ipswich Hospital NHS Trust, Ipswich, Suffolk
  - Northumbria Healthcare NHS Foundation Trust, North Shields, Tyne and Wear
  - Great Western Hospital NHS Foundation Trust, Swindon, Wiltshire
  - North Bristol NHS Trust - Southmead Hospital, Bristol
  - University Hospital of South Manchester NHS Trust, Manchester
  - Pennine Acute Hospitals NHS Trust, Manchester
  - South Tyneside NHS Foundation Trust, South Shields
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Hollen PJ, Gralla RJ, Liepa AM, Symanowski JT, Rusthoven JJ. Adapting the Lung Cancer Symptom Scale (LCSS) to mesothelioma: using the LCSS-Meso conceptual model for validation. Cancer. 2004 Aug 1;101(3):587-95. doi: 10.1002/cncr.20315. PMID 15274072
- [Background] Hollen PJ, Gralla RJ, Liepa AM, Symanowski JT, Rusthoven JJ. Measuring quality of life in patients with pleural mesothelioma using a modified version of the Lung Cancer Symptom Scale (LCSS): psychometric properties of the LCSS-Meso. Support Care Cancer. 2006 Jan;14(1):11-21. doi: 10.1007/s00520-005-0837-0. Epub 2005 Jul 6. PMID 15999264
- [Background] Langendijk H, Aaronson NK, de Jong JM, ten Velde GP, Muller MJ, Wouters M. The prognostic impact of quality of life assessed with the EORTC QLQ-C30 in inoperable non-small cell lung carcinoma treated with radiotherapy. Radiother Oncol. 2000 Apr;55(1):19-25. doi: 10.1016/s0167-8140(00)00158-4. PMID 10788684
- [Background] Montazeri A, Milroy R, Hole D, McEwen J, Gillis CR. Quality of life in lung cancer patients: as an important prognostic factor. Lung Cancer. 2001 Feb-Mar;31(2-3):233-40. doi: 10.1016/s0169-5002(00)00179-3. PMID 11165402